CLINICAL TRIAL: NCT02036489
Title: Pethema LAL-RI/2008: Treatment for Patients With Standard Risk Acute
Brief Title: Pethema LAL-RI/2008: Treatment for Patients With Standard Risk Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL-RI/2008
Record Dates: First submitted 2014-01-10; First posted 2014-01-15 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Acute Lymphobkastic Leukemia
MeSH Terms: interventions — Vincristine; Daunorubicin; Prednisone; Asparaginase; Cytarabine; Mercaptopurine; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Induction and consolidation treatment (Experimental)
  Interventions: Drug: Vincristine; Drug: Daunorubicin; Drug: Prednisone; Drug: L-asparaginase; Drug: Ciclophosphamide; Drug: Metotrexate; Drug: ARA-C; Drug: Hidrocortisone; Drug: Mercaptopurine; Drug: VP-16; Drug: Dexametasone

INTERVENTIONS:
Drug: Vincristine
Drug: Daunorubicin
Drug: Prednisone
Drug: L-asparaginase
Drug: Ciclophosphamide
Drug: Metotrexate
Drug: ARA-C
Drug: Hidrocortisone
Drug: Mercaptopurine
Drug: VP-16
Drug: Dexametasone

SUMMARY:
Understand the dynamics of elimination of MRD in adult patients with standard-risk LAL treated with a pediatric protocol.

DETAILED DESCRIPTION:
Induction therapy is administered. Patients experiencing slow response (> 10 % blasts in the 15th mo of treatment) were included in the LAL -AR -03 protocol, on the arm of intensified induction. Those who do not reach the RC will be excluded from the study and will be treated according to the protocol LAL-AR/03 , which will be incorporated receiving blocks consolidation. All patients in CR consolidation treatment (1 and 2 ) followed reinducciones maintenance (maintenance -1 ) to complete the first year of treatment and maintenance without reinducciones (maintenance -2 ) to complete two years from the RC will be administered . If after union persistent high levels of ER ( > 0.05 %) and this reappears later during maintenance therapy the patient will be excluded from the study and will be treated according to the protocol of high risk ( PETHEMA LAL-AR/03 ) . In case of persistent high levels of ER patients after consolidation will consolidate blocks PETHEMA LAL-AR/03 protocol followed by allogeneic HSCT . If the ER reappears during maintenance treatment the patient will receive an allogeneic HSCT , Standby thereof, may be administered one or two blocks consolidation of LAL -AR -03 protocol.

To allow time to better characterize the LLA and thus ensure proper inclusion of patients in the study recommends administering a prephase with :

- Prednisone ( PDN) 60 mg/m2 po or iv through characterization of LAL with a maximum of 7 days.

intrathecal chemotherapy

* Methotrexate (MTX ) : 12 mg
* ARA - C: 30 mg
* Hydrocortisone 20 mg

The LAL meeting the inclusion criteria, the study may continue

Induction chemotherapy

* Vincristine (VCR ) 1.5 mg/m2 ( maximum dose 2 mg ) iv on days 1 and 8.
* daunorubicin (DNR ) 30 mg/m2 iv on days 1 and 8.
* Prednisone ( PDN ): 60 mg/m2 night , i.v. or p.o , 1-14 days

Study of bone marrow at day +14

* Less than 10% blasts ( by morphology) or hypocellular bone marrow
* Vincristine (VCR ) 1.5 mg/m2 ( maximum dose 2 mg) iv 15 and 22
* daunorubicin (DNR ) 30 mg/m2 i.v 15 and 22
* L -asparaginase ( L -ASA ) of E. coli ( Kidrolase ® ) : 10,000 IU/m2 , iv , 16-20 , 23-27 .
* 1,000 mg/m2 cyclophosphamide , i.v. day 36
* Prednisone ( PDN) :
* 60 mg/m2 per day, i.v or p.o , days 15-27
* 30 mg/m2 per day, i.v or p.o , days 28-35
* Equal to or more than 10 % blasts ( by morphology)
* Step PETHEMA protocol LAL-AR/2003

Intrathecal chemotherapy

* Methotrexate (MTX ) 12 mg days 1 and 29
* ARA- C: 30 mg days 1 and 29
* Hydrocortisone 20 mg days 1 and 29

Evaluation at the end of induction (day 28 or when a finding hemoperiférica recovery)

* Patients RC : consolidation -1
* Patients without RC : excluded. Step PETHEMA LAL-AR/2003 protocol .

Study of the ER at the end of induction. Molecular response was considered if the ER is < 0.01 %. Although a molecular response is not achieved , the patient will remain in the protocol if you have standard response at day 14 and is in CR at day 28 .

Consolidation treatment -1 These cycles include known cytostatics LAL activity against at intermediate or high doses. This phase of treatment as possible to begin two weeks of the administration of the last dose of cytostatic induction phase . The patient should have a WBC count > 3x109 / L (granulocytes > 1.5 x 109 / L ) and platelets > 100x109 / L.

Mercaptopurine ( MP ) 50 mg/m2 , po, days 1-7 , 28-35 and 56-63 MTX : 3 g/m2 iv , in 24 hours , day 1, 28 and 56 . For administration, and rescue treatment should be followed the rules specified below .

VP -16 100 mg/m2 ( infusion 1 hour), 14-15 and 42-43 ARA- C 500 mg/m2 iv every 12 hours , 3 hours , 14-15 and 42-43 . Intrathecal Chemotherapy or Methotrexate ( MTX ) 12 mg on days 1, 28 and 56 or ARA- C: 30 mg days 1, 28 and 56 or Hydrocortisone 20 mg days 1, 28 and 56

Treatment consolidation-2/reinduction It consists of a cycle similar to the induction chemotherapy . It will start if possible within one week of completion of the last dose of mercaptopurine in the previous cycle (thus, from the 18th week of the start of treatment) .

Dexamethasone (DXM ) :

or 10 mg/m2 per day, p.o or i.v 1-14 days to 5 mg/m2 night , p.o or i.v., day 15 to 21 VCR 1.5 mg/m2 , i.v. , days 1, 8 and 15 DNR : 30 mg/m2 , i.v. , 1, 2 , 8 and 9 CFM and 600 mg/m2 day , i.v. , days 1 and 15 L -ASA E. coli ( Kidrolase ® ) : 10,000 IU/m2 i.m. or i.v., on days 1-4 and 15-18 .

Intrathecal Chemotherapy or methotrexate (MTX ) 12 mg days 1 and 15 or ARA- C: 30 mg days 1 and 15 or Hydrocortisone 20 mg days 1 and 15

Evaluation of ER at the end of the consolidation A cytofluorometric study fee is mo If the ER is > 0.05 % (tested on two separate occasions 15 days ) the patient will go to high-risk protocol ( PETHEMA LAL-AR/2003 ) .

If ER < 0.05 % the patient continue the protocol.

Maintenance treatment with 1 reinducciones It will consist of continuous administration of chemotherapy ( mercaptopurine and methotrexate ) with reinducciones up to a year from the start of treatment. It lasts therefore between approximately 22 and 52 weeks of treatment.

Continuous Chemotherapy

* MP 50 mg/m2 per day, p.o
* MTX 20 mg/m2 per week , i.m. Reinducciones
* VCR 1.5 mg/m2 ( maximum dose 2 mg) , iv , day 1.
* PDN 60 mg/m2 night , i.v. or p.o , days 1-7
* L - ASA E. coli ( Kidrolase ® ) : 20,000 IU/m2 i.m. or i.v. , day 1.
* Intrathecal Chemotherapy Methotrexate (MTX ) 12 mg 1st ARA- C: 30 mg 1st Hydrocortisone 20 mg Day 1

During the week of administration of each cycle of chemotherapy reinduction continuous suspended.

Evaluation after the fourth reinduction . Immunophenotypic study of a new bone marrow will be made

* If ER is < 0.01 % , subsequent reinducciones are suspended and continues only with continuous chemotherapy until week 52 , at which point it switches to maintenance -2.
* If ER between 0.05% and 0.01% , the reinducciones 5 was administered to 8
* If ER > 0.05 % (tested on two separate occasions 15 days ) the patient will go to high-risk protocol ( PETHEMA LAL-AR/2003 ) .

Treatment Support 2 It consisitirá in continuous administration of chemotherapy ( mercaptopurine, and methotrexate ) to complete two years in continuous complete remission .

* MP 50 mg/m2 per day, p.o
* MTX 20 mg/m2 per week , i.m. Throughout the maintenance treatment should seek to retain WBC counts between 2.5 and 5x109 / L and platelet counts above 120x109 / L. If these lower limits should be reduced is decreased by 20 % doses of MP and MTX. If the numbers of leukocytes exceed 5x109 / L will increase by 20 % the dose of MP (50 to 60 mg/m2 )

ELIGIBILITY:
Inclusion Criteria:

Adults (age> 15 years) with ALL standard risk previously untreated. The LAL standard risk is defined by all of the following criteria:

* Age less than 30 years
* WBC <25x109 / L
* Absence of cytogenetic alterations that misbehave forecast or t (9, 22) or demonstration of BCR-ABL rearrangement or alterations in 11q23, or demonstration ALL1-AF4 rearrangement (MLL)

Exclusion Criteria:

LAL L3 type mature phenotype B (sIg +) or with cytogenetic abnormalities characteristic of Burkitt LAL (t [8, 14], t [2, 8], t [8, 22]). For these patients have the BURKIMAB study.

* LAL Ph (BCR-ABL) positive. These patients should be treated with imatinib associated with chemotherapy.
* Biphenotypic acute leukemias and bilinear. For these patients treatment is recommended LAM own guidelines.
* Acute undifferentiated leukemias. For these patients treatment is recommended LAM own guidelines.
* Patients with a history of coronary artery disease, valvular or hypertensive heart disease.
* Patients with chronic liver disease.
* Patients with chronic respiratory failure.
* Renal failure not due to the LAL.
* Severe neurological disorders, not due to the LAL.
* General State concerned (grades 3 and 4 WHO scale), not attributable to the LAL.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of treatment in adulta with standard risk acute lymphoblastic leukemia | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Germans Trias i Pujol, Barcelona, Spain